CLINICAL TRIAL: NCT05932979
Title: Effect of the Administration of L-arginine vs. Placebo on the vHIT Result, Vestibular Caloric Tests and Symptoms of Patients Diagnosed With Presbyvestibulopathy.
Brief Title: Effect of the Administration of L-arginine vs. Placebo in Patients Diagnosed With Presbyvestibulopathy.
Acronym: L-ARGPRES
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the investigation was cancelled because there was no monetary resource to complete it.
Sponsor: Centro Universitario de Tonalá (Other)
Responsible Party: Principal Investigator, Martha De Nuestra Señora De San Juan Rodríguez Sahagún, Investigator, Centro Universitario de Tonalá
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 160/22
Record Dates: First submitted 2023-05-12; First posted 2023-07-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Presbyvestibulopathy
Keywords: L-arginine; Presbyvestibulopathy; Vertigo; v-HIT
MeSH Terms: conditions — Vertigo | interventions — Arginine; Starch

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical trial with a placebo control group.
Who Masked: Participant, Investigator
Masking Description: Patients will be assigned by simple randomization using a table of random numbers to the pharmacological intervention groups.
  The study treatment and treatment assignment codes will be kept in custody by someone outside the research team. In addition, it will be in charge of the delivery, reception and meticulous counting of the capsules to guarantee the blindness and adherence to the treatment by the patients.
  This study is considered double-blind since both the principal investigator and the patient are unaware of the pharmacological intervention to which the patients will be assigned. Blinding will be possible thanks to the homologation of the drug and the placebo in both groups with capsules identical in shape, size and colour. In the same way, the medicine will be delivered in bottles of the same size, shape and color, identified only with the allocation code.
  The blind may be broken in the presence of serious adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-arginine (Experimental): L-arginine 3 grams per day, divided into doses of 1 g every 8 hours during 90 days.
  Interventions: Drug: L-arginine
- Placebo (Placebo Comparator): Starch 1 gr every 8hr, during 90 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-arginine — L-arginine 2-amino-5-guanidino-pentanoic acid is a proteinogenic amino acid that is a natural constituent of the protein diet.
  Other Names: Arginine
  Arms: L-arginine
Other: Placebo — Starch
  Other Names: Starch
  Arms: Placebo

SUMMARY:
Presbivestibulopathy is defined as a chronic vestibular syndrome characterized by bilateral vestibulopathy verified with vestibular tests. These tests objectively assess vestibular function: video Head Impulse Test (v-HIT) and Vestibular Caloric Tests. Also, there are some questionnaires that serve us for monitoring and prognosis (Dizziness Handicap Inventory). There is currently no specific treatment for presbyvestibulopathy. The objective of this study is to evaluate the effect of L-arginine vs. placebo on symptoms, changes in the results of vHIT tests of patients diagnosed with presbyvestibulopathy. It will be conducted a randomized, double blind, placebo controled clinical trial. Patients will be men and women who meet the diagnostic criteria for Presbyvestibulopathy of the Barany Society. The sample size will be 12 patients per group. The patients in the experimental group will receive L-arginine at a dose of 3 grams divided into three doses of 1 g (capsules) every 8 hours, for 3 months. Patients in the control group will receive placebo at the same dosage. All patients will receive vestibular rehabilitation exercises. At the beginning and the end of the intervention , the following tests will be carried out: vertigo disability questionnaire, vHIT tests, and the Up and Go time test.

DETAILED DESCRIPTION:
Vertigo is a common cause in the otorhinolaryngology consultation; a high incidence of this condition has been reported, since there are reports indicating that up to 80% of the world population has presented an episode of vertigo at some stage of their lives.

In Germany, it has been reported a prevalence of moderate to severe vestibular vertigo is reported, calculated using a representative sample of a 22.9% in adults of 18 to 79 years. In a report of the United States Emergency Department, it has been reported that 3.3% of the first-contact consultations are due to dizziness, of which 32.9% wer of otological or vestibular origin.

Vertigo is classified into two categories: vertigo of central origin and peripheral vertigo. Peripheral vertigo, object of study of this investigation, is originated in the vestibular system, located in the inner ear. Among the differential diagnoses of vertigo of peripheral origin we find presbivestibulopathy, which is a condition characterized by bilateral vestibular dysfunction proven with objective diagnostic tests such as video HIT (vHIT), vestibular caloric tests, among others. In addition, the diagnostic must be done in people over 60 years, and other diagnostic criteria established by the diagnostic criteria for Presbyvestibulopathy of the Barany Society.

The treatment of vertigo, as well of the presbyvestibulopathy, is aimed to stabilize the pathological fluctuations in peripheral vestibular function, as well as promoting central compensation in case of a permanent deficit in vestibular function. Therefore, the drugs used for its treatment their purpose is to regulate the decompensated vestibular activity and to improve the symptoms, but not to suppress the cause that originates the pathology since the mechanism of action of the disease is not well established.

Currently, there is not a first-choice medication for the treatment of vertigo in general, much less for presbyvestibulopathy, since none has show high efficacy and low presence of adverse effects.

Some of the drugs used to treat vertigo include anticholinergics, antihistamines, benzodiazepines and calcium channel blockers.

In the same way, some substances have been used that have shown effectiveness despite the fact that their mechanism of action is unknown or not very clear, sus as betahistine and Gingko biloba.

L-arginine is a precursor amino acid fr the endogenous synthesis of nitric oxide (NO), a molecule produced in the vascular endothelium with vasodilatory, antiatherogenic and antiplatelet action.

To date, there is no evidence of the use of L-arginine for the treatment of vertigo, however, its vasodilator effect as a precursor of NO should favor vascular perfusion in the vestibular system, therefore, it is of interest to know the therapeutic effects of L-arginine for ths treatment of pathology.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Age over 60 years.
* That patient meets the diagnostic criteria established for presbyvestibulopathy by the Classification Committee of the Barany Society:

  * Chronic vestibular syndrome (al least 3 months duration) with at least 2 of the following symptoms:

    * Postural imbalance or unsteadiness
    * Gait disturbance
    * Chronic dizziness
    * Recurrent falls
  * Mild bilateral peripheral vestibular hypofunction documented by at leat 1 of the following:

    * VOR gain measured by video-HIT between 0.6 and 0.8 bilaterally
    * VOR gain between 0.1 and 0.3 upon sinusoidal stimulation on a rotatory chair (0.1 Hz, Vmax=50-60°/sec)
    * Reduced caloric response (sum of bithermal saccadic peak velocity (SPV) on each side between 6 and 25°/sec)
  * Age ≥60 years
  * Not better accounted for by another disease or disorder
* Consent under information

Exclusion Criteria:

* Not being able to rule out the use of antivertigo drugs 1 week prior to study entry.
* Use of vasodilator drugs or antihistamines.
* Orthostatic hypotension
* Cognitive deficit of the patient that prevents him from understanding the implications of the study.
* Known uncontrolled liver or kidney disease.
* Known hypersensitivity to study drugs.
* Chronic use of drugs with an anticoagulant effect.
* Bronchial asthma.

Elimination Criteria:

* Treatment adherence <80% evaluated through registration in an adherence diary and capsules count
* Presence of serious adverse events
* Withdrawal of consent under information

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Baseline Video Head Impulse Test vHIT | Pre-intervention
  The vHIT is a simple, rapid test to assess vestibular function. It is based on the physiological aspects of the vestibular ocular reflex (VOR). VOR is a rapid reflex with a duration of 7 to 10 milliseconds and consists of the ability to keep the gaze fixed on an object with rapid and unexpected movements of the head.
  This study has a specificity and sensitivity of 100% to evaluate the VOR.
Final Video Head Impulse Test vHIT | Final (after 90 days of intervention)
  The vHIT is a simple, rapid test to assess vestibular function. It is based on the physiological aspects of the vestibular ocular reflex (VOR). VOR is a rapid reflex with a duration of 7 to 10 milliseconds and consists of the ability to keep the gaze fixed on an object with rapid and unexpected movements of the head.
  This study has a specificity and sensitivity of 100% to evaluate the VOR.
Baseline Dizziness Handicap Inventory | Pre-intervention
  Questionnaire that helps us to know the degree of emotional, functional and physical disability of patients diagnosed with presbyvestibulopathy. In addition, it has been used by different authors as a prognostic value, to know the improvement of pre- and post-treatment patients.
Final Dizziness Handicap Inventory | Final (after 90 days of intervention)
  Questionnaire that helps us to know the degree of emotional, functional and physical disability of patients diagnosed with presbyvestibulopathy. In addition, it has been used by different authors as a prognostic value, to know the improvement of pre- and post-treatment patients.

SECONDARY OUTCOMES:
Baseline Time up and go Test | Pre-intervention
  It is a simple test that consists of a patient being asked to stand up without support while sitting in a chair without armrests and walk forward for 3 meters and back, the time it takes to do so is timed. Most authors consider that if the duration is greater than 10 seconds, there is a greater risk of falls.
Final Time up and go Test | Final (after 90 days of intervention)
  It is a simple test that consists of a patient being asked to stand up without support while sitting in a chair without armrests and walk forward for 3 meters and back, the time it takes to do so is timed. Most authors consider that if the duration is greater than 10 seconds, there is a greater risk of falls.
Adverse events | Final (after 90 days of intervention)
  Adverse events will be evaluated through a diary in which patients will record any adverse event presented between visits. Also, it will be verified with direct interview.
Initial Audiometry | Pre-intervention
  Audiometry aims to make a graphic record of hearing which is called audiogram. This study help us to detect hearing loss and classiffy it according to its site of origin.
Final Audiometry | Final (after 90 days of intervention)
  Audiometry aims to make a graphic record of hearing which is called audiogram. This study help us to detect hearing loss and classiffy it according to its site of origin.

CONTACTS AND LOCATIONS:
Overall Officials: Martha de Nuestra Señora de San Juan Rodríguez, MD, Principal Investigator — CUTonalá
Locations (1):
- CUTonalá, Tonalá, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agrawal Y, Van de Berg R, Wuyts F, Walther L, Magnusson M, Oh E, Sharpe M, Strupp M. Presbyvestibulopathy: Diagnostic criteria Consensus document of the classification committee of the Barany Society. J Vestib Res. 2019;29(4):161-170. doi: 10.3233/VES-190672. PMID 31306146
- [Background] Aggarwal NT, Bennett DA, Bienias JL, Mendes de Leon CF, Morris MC, Evans DA. The prevalence of dizziness and its association with functional disability in a biracial community population. J Gerontol A Biol Sci Med Sci. 2000 May;55(5):M288-92. doi: 10.1093/gerona/55.5.m288. PMID 10819319
- [Background] Alrwaily M, Whitney SL. Vestibular rehabilitation of older adults with dizziness. Otolaryngol Clin North Am. 2011 Apr;44(2):473-96, x. doi: 10.1016/j.otc.2011.01.015. PMID 21474018
- [Background] Bai Y, Sun L, Yang T, Sun K, Chen J, Hui R. Increase in fasting vascular endothelial function after short-term oral L-arginine is effective when baseline flow-mediated dilation is low: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2009 Jan;89(1):77-84. doi: 10.3945/ajcn.2008.26544. Epub 2008 Dec 3. PMID 19056561
- [Background] Rodrigues DL, Ledesma ALL, Pires de Oliveira CA, Bahmad F Jr. Effect of Vestibular Exercises Associated With Repositioning Maneuvers in Patients With Benign Paroxysmal Positional Vertigo: A Randomized Controlled Clinical Trial. Otol Neurotol. 2019 Sep;40(8):e824-e829. doi: 10.1097/MAO.0000000000002324. PMID 31356483
- [Background] Dong JY, Qin LQ, Zhang Z, Zhao Y, Wang J, Arigoni F, Zhang W. Effect of oral L-arginine supplementation on blood pressure: a meta-analysis of randomized, double-blind, placebo-controlled trials. Am Heart J. 2011 Dec;162(6):959-65. doi: 10.1016/j.ahj.2011.09.012. Epub 2011 Nov 8. PMID 22137067
- [Background] Rosengren SM, Young AS, Taylor RL, Welgampola MS. Vestibular function testing in the 21st century: video head impulse test, vestibular evoked myogenic potential, video nystagmography; which tests will provide answers? Curr Opin Neurol. 2022 Feb 1;35(1):64-74. doi: 10.1097/WCO.0000000000001023. PMID 34889807
- [Background] Scholtz AW, Hahn A, Stefflova B, Medzhidieva D, Ryazantsev SV, Paschinin A, Kunelskaya N, Schumacher K, Weisshaar G. Efficacy and Safety of a Fixed Combination of Cinnarizine 20 mg and Dimenhydrinate 40 mg vs Betahistine Dihydrochloride 16 mg in Patients with Peripheral Vestibular Vertigo: A Prospective, Multinational, Multicenter, Double-Blind, Randomized, Non-inferiority Clinical Trial. Clin Drug Investig. 2019 Nov;39(11):1045-1056. doi: 10.1007/s40261-019-00858-6. PMID 31571128
- [Background] Sokolova L, Hoerr R, Mishchenko T. Treatment of Vertigo: A Randomized, Double-Blind Trial Comparing Efficacy and Safety of Ginkgo biloba Extract EGb 761 and Betahistine. Int J Otolaryngol. 2014;2014:682439. doi: 10.1155/2014/682439. Epub 2014 Jun 25. PMID 25057270
- [Background] Agrawal Y, Zuniga MG, Davalos-Bichara M, Schubert MC, Walston JD, Hughes J, Carey JP. Decline in semicircular canal and otolith function with age. Otol Neurotol. 2012 Jul;33(5):832-9. doi: 10.1097/MAO.0b013e3182545061. PMID 22699991